CLINICAL TRIAL: NCT04608214
Title: Evaluation of the Efficacy, Safety and Tolerability of Alisporivir for the Treatment of Hospitalised Patients With Infections Due to SARS-CoV-2 (COVID-19). A Randomised, Open-label, Proof of Concept, Phase 2 Study
Brief Title: Evaluation of Alisporivir for the Treatment of Hospitalised Patients With Infections Due to SARS-CoV-2 (COVID-19)
Acronym: CYCLOVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200552; 2020-002295-13 (Other: N° IDRCB)
Record Dates: First submitted 2020-10-12; First posted 2020-10-29 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2
Keywords: Alisporivir; Viral Load; efficacy; safety; tolerability
MeSH Terms: interventions — alisporivir; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomised, open-label, proof of-concept, Phase 2 study to evaluate the efficacy, safety and tolerability of alisporivir plus SOC as compared to SOC for the treatment of hospitalised patients with infections due to SARS-CoV-2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alisporivir (Experimental): Administration of alisporivir and standard of care (SOC)
  Interventions: Drug: Alisporivir
- Standard of care (SOC) (Active Comparator): Locally accepted regimen protocols for patient care
  Interventions: Other: Standard of care (SOC)

INTERVENTIONS:
Drug: Alisporivir — Administration of alisporivir at the dose of 600 mg p.o. BID from D1 to D14 to patients and standard of care (SOC).
  Arms: Alisporivir
Other: Standard of care (SOC) — Locally accepted regimen protocols for patient care and select agents based on the underlying diagnosis and the severity of COVID 19 (excepting e.g. azithromycin and other antibiotics listed as prohibited medications)
  Arms: Standard of care (SOC)

SUMMARY:
COVID-19 is a viral respiratory and systemic disease that has been rapidly spreading globally since the first cases were reported in December 2019 and has now become pandemic. The causative agent of COVID-19 was identified as a novel coronavirus named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2, first designated as 2019-nCoV).

The disease manifestations of COVID-19 can range from mild, self-resolving respiratory disease to severe pneumonia, ARDS, multiorgan failure, and ultimately death. In early reports, the mortality rate among patients admitted to hospital and with confirmed SARS-CoV-2 infection was reported to be between 4 and 15%. Although the disease can afflict all age groups, elderly patients and patients with underlying comorbidities such as high body mass index, hypertension, diabetes, cardiovascular disease, or cerebrovascular disease are at risk of developing severe disease and dying.

There are currently no etiologic treatments for COVID-19, and efforts are underway to identify therapeutics that could be effective in controlling this disease.

DETAILED DESCRIPTION:
Cyclophilins are cellular (host) peptidyl-prolyl cis/trans isomerases (molecular chaperones) involved in protein folding, maturation, and trafficking. Cyclophilins have been shown to play a key role in the lifecycle of many coronaviruses, including human coronaviruses 229E (HCoV-229E) and NL-63 (HCoV-NL63), feline infectious peritonitis coronavirus (FPIV), SARS-CoV and Middle-East-Respiratory-Syndrome coronavirus (MERS-CoV). Cyclosporin A (CsA), a potent cyclophilin inhibitor, blocks the replication of various coronaviruses in vitro, including HCoV-229E, HCoV-NL63, FPIV, mouse hepatitis virus (MHV), avian infectious bronchitis virus, and SARS-CoV.

Alisporivir is a non-immunosuppressive analogue of CsA with potent cyclophilin inhibition properties. In vitro, alisporivir inhibits the replication of HCoV-229E, HCoV-NL63, MHV, SARS-CoV and MERS-CoV at low micromolar concentrations without cytotoxic effect. Although alisporivir has not demonstrated activity against coronaviruses in in vivo models to date, recent experiments showed that alisporivir bears concentration-dependent properties against CoV-2 in vitro.

Preclinical pharmacology data indicate that, after oral administration, alisporivir is widely distributed in the whole body, including the lungs. Furthermore, the EC90 of alisporivir against SARS-CoV-2 in VeroE6 cells appears to be clinically achievable in patients. In addition, because alisporivir inhibits all cellular cyclophilins, it also blocks mitochondrial cyclophilin-D, a key regulator of mitochondrial permeability transition pore (mPTP) opening, a mechanism involved in triggering cell death.

Therefore, besides its antiviral properties, alisporivir may also be effective in preventing lung tissue damage.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females ≥18 years and ≤80 years of age at the time of screening.
2. Are hospitalised during the screening period with duration of hospitalisation prior to randomisation ≤48 hours.
3. Have a diagnosis of COVID-19 based on symptoms onset and positive SARS-CoV-2 RT-PCR test from nasopharyngeal swab.
4. Viral load ≤ 30 Ct
5. Have at least one (1) of the following:

   1. Radiographic pulmonary infiltrates (CT scan), AND/OR
   2. Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤94% on room air, AND/OR
   3. Requirement for supplemental oxygen.
6. If female, of non-childbearing potential or if of childbearing potential, be willing to commit to either sexual abstinence or use of at least 2 medically accepted, effective methods of birth control from screening through 2 months after last alisporivir dose.
7. If male, a willingness to refrain from donating sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective method of birth control from screening through 4 months after last alisporivir dose.
8. Willing and able to provide written informed consent.
9. Willing to comply with all study assessments and adhere to the protocol schedule.
10. Has an affiliation with a social security system.

Exclusion Criteria:

1. Patients requiring mechanical ventilation at screening or randomisation.
2. In the opinion of the investigator, the patient is unlikely to survive the following 7 days after randomisation due to a rapidly progressive or terminal illness with a high risk of mortality due to any cause, including acute hepatic failure, respiratory failure or severe septic shock.
3. Patients who are unconscious or considered by the investigator unable to consent.
4. Other severe co-morbidity with life expectancy ≤3 months according to the investigator's assessment.
5. Critically ill patients who have an APACHE II score ≥30.
6. Concomitant severe bacterial infection including blood stream infections, endocarditis, osteomyelitis, retroperitoneal abscess, septic arthritis, or meningitis diagnosed within 7 days prior to randomisation (bacterial pulmonary infection that may complicate COVID-19 is not an exclusion criterion).
7. Any of the following signs of severe sepsis:

   1. Shock or profound hypotension defined as systolic blood pressure ≤90 mm Hg or a decrease of ≥40 mm Hg from the value obtained during screening that is not responsive to fluid challenge.
   2. Hypothermia (core temperature ≤ 35.6°C).
   3. Disseminated intravascular coagulation (DIC) as evidenced by PT, PTT 2 × upper limit of normal (ULN), or platelets ≤ 50% of the lower limit of normal (LLN).
8. History of positive test for human immunodeficiency virus (HIV) including all patients currently on highly active antiretroviral therapy (HAART) regardless of the CD4+ cell count.
9. Presence of immunodeficiency or an immunocompromised condition including neutropenia, haematologic malignancy, history of haematopoietic stem cell transplant, history of solid organ transplant, receiving immunosuppressive therapy and long term use of systemic corticosteroids.
10. Severe hepatic impairment at screening, as evidenced by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 5 × ULN or total bilirubin ≥2 × ULN (except in case of known Gilbert syndrome), or clinical signs of decompensated cirrhosis or end-stage hepatic disease (e.g., ascites, hepatic encephalopathy).
11. Acute hepatitis, decompensated cirrhosis (any Child-Pugh B or C class), acute hepatic failure or acute decompensation of chronic hepatic failure.
12. Severe renal impairment (creatinine-clearance ≤30 mL/min) or end-stage renal disease (ESRD) requiring haemodialysis or peritoneal dialysis, according to Cockcroft-Gault.
13. Uncontrolled hypertension that is not responsive to treatment.
14. Uncontrolled thyroid function (Thyroid Stimulating Hormone [TSH] outside of normal ranges).
15. History of epilepsy or known seizure disorder (excluding a history of childhood febrile seizures).
16. Acute co-morbidity within 7 days before inclusion such as myocardial infarction.
17. A female who is pregnant or breastfeeding.
18. Documented hypersensitivity reaction or anaphylaxis to alisporivir, one of the non-active ingredients or any of the SOC medications.
19. Receipt of any investigational medication in the 3 months prior to screening.
20. Anticipated transfer to another hospital that is not a study site during the first 4 days of treatment.
21. Patients previously treated with antivirals, immunomodulators (mAbs in the 3 months prior to screening) and other medicines prohibited in this study in the 14 days prior to randomisation.
22. Ongoing or recent use of any other medication (including over the counter medication and herbal products) within 14 days before randomisation or within 5 drug half-lives of that medication (whichever is longer) that are known inhibitors/inducers of cytochrome P450 3A or P-glycoprotein (P-gp), or inhibitors of organic anion transporting polypeptides (OATPs), multi resistance protein 2 (MRP2) or bile salt export pump (BSEP).

    Known need of concomitant treatment with the following medications during treatment with alisporivir and 14 days after the end of treatment:
    1. Known inhibitors/inducers of cytochrome P450 3A or P-gp, or inhibitors of OATPs, MRP2 or BSEP;
    2. Drugs with narrow therapeutic index that are known sensitive substrates of cytochrome P450 3A, or substrates of P-gp, OATPs, MRP2 or BSEP.
23. Any other condition or prior therapy, which, in the opinion of the investigator, would make the patient unsuitable for this study.
24. Patients with history of pancreatic disease.
25. Patients under legal protection.
26. Prisoners.
27. Patients participating in another interventional study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 viral load in nasopharyngeal swabs | at Day 1 and Day 7

SECONDARY OUTCOMES:
Viral Load Response Rate (VLRR) | at Day 1 and Day 7
Percentage of patients reporting each severity rating on an 8-point ordinal scale. | at Day 1, Day4, Day 7, Day 11, Day 14 and Day 90
Change in National Early Warning Score scale | at Day 1, Day 4, Day 7, Day 11, Day 14 and Day 90
Changes in thoracic CT scan | screening to Day 1, Day 14 and Day 90
Percentage of patients admitted to Intensive Care Unit (ICU) | at Day 1 to Day 28
Time to admission to Intensive Care Unit (ICU) | at Day 1 to Day 28
Percentage of patients admitted to Intensive Care Unit (ICU) | at Day 90
Time to admission to Intensive Care Unit (ICU) | at Day 90
Percentage of patients requiring mechanical ventilation | at Day 1 to Day 28
Percentage of patients requiring mechanical ventilation | at Day 90
Percentages of patients negative for SARS CoV 2 RNA in nasopharyngeal swabs | at Day 14, Day 21 and Day 28
Time to negative viral load | at Day 1 to Day 28
Time to resolution of symptoms | at Day 1 to Day 28
Time to resolution of symptoms | at Day 90
Duration of need for supplemental oxygen | at Day 1 to Day 28
Duration of need for supplemental oxygen | at Day 90
Duration of hospitalisation | at Day 1 to Day 28
Duration of hospitalisation | at Day 90
Duration of new non-invasive ventilation or high flow oxygen use | at Day 1 to Day 28
Duration of new non-invasive ventilation or high flow oxygen use | at Day 90
Duration of new oxygen use | at Day 1 to Day 28
Duration of new oxygen use | at Day 90
Duration of new ventilator or ECMO use | at Day 1 to Day 28
Duration of new ventilator or ECMO use | at Day 90
Number of non-invasive ventilation/high flow oxygen free days | at Day 1 to Day 28
Number of non-invasive ventilation/high flow oxygen free days | at Day 90
Number of oxygenation free days | at Day 1 to Day 28
Number of oxygenation free days | at Day 90
Patient all-cause mortality | at Day 14, Day 28 and Day 90
Cumulative incidence of any AE | at Day 1 to Day 90
Cumulative incidence of Grade 3 and 4 AEs | at Day 1 to Day 90
Cumulative incidence of SAEs | at Day 1 to Day 90
Percentage of re-hospitalization | Hospital discharge to D90 ±2d

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel PAWLOTSKY, MD, PhD, Study Director — Assistance Publique Hôpitaux de Paris (AP-HP)
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU Henri Mondor, Créteil, France